CLINICAL TRIAL: NCT04408001
Title: Study of Kinetics and Efficacy of the Immune Response Against COVID-19 Among Hospital Staff
Acronym: IMMUNO-COVID
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-04; 2020-A01019-30 (Other: IDRCB)
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples ans saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic individuals: Hospital staff identified by the COVID-19 case census cell :
  * who have been infected (confirmed by a positive RT-PCR result on a nasopharyngeal swab)
  * OR who have displayed clinical signs compatible with COVID-19 despite a negative RT-PCR result.
  Interventions: Other: Clinical interview; Biological: Blood collection; Biological: Saliva collection
- Asymptomatic individuals: Hospital staff who have not been identified by the COVID-19 case census cell.
  Interventions: Other: Clinical interview; Biological: Blood collection; Biological: Saliva collection

INTERVENTIONS:
Other: Clinical interview — At each study visit, participants will be questioned by a physician about their persistent symptoms or the existence of intercurrent infections that may resemble COVID-19.
Biological: Blood collection — At each study visit,
  * 1 EDTA tube for complete blood count
  * 3 dry tubes with gel for serology, serum neutralisation test and serum library
  * 1 cell preparation tube for the separation of immune cells within the circulating blood will be collected.
Biological: Saliva collection — At each study visit, a saliva sample will be collected for the determination of IgA antibodies.

SUMMARY:
COVID-19 is a pathology linked to the SARS-CoV-2 virus, a new virus of the coronaviridae family that emerged in China in December 2019 before rapidly becoming a pandemic according to the WHO on March 11, 2020. The epidemic affected France from February 2020. On February 24, a patient hospitalized at Percy hospital was the cause of a major nosocomial epidemic, potentially responsible for more than 250 symptomatic people in the hospital as of April 6. The outbreak was identified by Percy hospital management on March 16, and barrier measures were immediately put in place. From March 20, a mixed investigation unit set up a chain of nasopharyngeal swabs for Percy hospital staff.

A COVID-19 case reporting unit was set up at Percy hospital in response to the identification of the outbreak within the hospital. This unit carried out rapid identification and regular follow-up until the return to work of the staff. Thus all symptomatic patients are identified and the COVID-19 case census cell will follow all Percy hospital staff, including volunteers recruited to deal with the epidemic, throughout the duration of the epidemic. This population, captive by nature, will be one of the few described in the world during this epidemic.

Current data on short-, medium- and long-term immunity induced by COVID-19 infection are fragmentary, as is the existence of a large asymptomatic population, making it difficult to cut the chains of transmission in the absence of an effective diagnostic tool.

Another important issue is the quality of immunity induced by the infection, as it conditions the future of the pandemic, which could become endemic and recurrent if immunity were not sterilizing. As yet unpublished data in primates show that in the primate model re-infection is not possible in the short term, while patients cured from the Wuhan epidemic seem to be detected again positive for virus shedding.

The objective of this study is to characterize the immunity (systemic and local) induced by SARS-Cov-2 infection among Percy hospital staff who are at high risk of contamination even in a period of confinement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Military or civilian or contactual volunteer on duty at Percy hospital during the COVID-19 pandemic.

Exclusion Criteria:

* Individuals who have displayed a severe form of early-onset COVID-19 who required intensive care management or hospitalization;
* Presence of factors modulating immunity with congenital or acquired immunosuppression:

  * Medication: cancer chemotherapy, immunosuppressive drugs, biotherapy, corticosteroids
  * Uncontrolled HIV infection or CD4 <200/mm3 infection
  * History of solid organ or hematopoietic stem cell transplants

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Percy hospital staff having (symptomatic individuals group) or not (asymptomatic individuals group) presented COVID-19 infection symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Induced SARS-CoV2 immunity | At day 21 (compared to enrollment [Day 0])
  The presence of induced immunity will be identified by an Ig family switch on the first two serologies with a high titre of specific IgG and disappearance of IgM.
Long-term protection of induced SARS-CoV2 immunity at 6 months | 6 months following enrollment
  The presence of induced immunity will be identified on serology analysis at 6 months.
Long-term protection of induced SARS-CoV2 immunity at 1 year | 1 year following enrollment
  The presence of induced immunity will be identified on serology analysis at 1 year.
Anti-SARS-CoV2 antibodies kinetics in blood throughout the study | From enrollment (Day 0) to 1 year after enrollement
  Kinetics of anti-SARS-CoV-2 antibodies using ELISA technique on serum samples from enrollment (Day 0) to 1 year after enrollement
Anti-SARS-CoV2 antibodies kinetics in saliva throughout the study | From enrollment (Day 0) to 1 year after enrollement
  Kinetics of anti-SARS-CoV-2 antibodies using ELISA technique on saliva samples from enrollment (Day 0) to 1 year after enrollement
Kinetics of serum neutralization in blood throughout the study | From enrollment (Day 0) to 1 year after enrollement
  Kinetics of serum neutralization against SARS-CoV-2 positive using ELISA technique on serum samples from enrollment (Day 0) to 1 year after enrollement.

SECONDARY OUTCOMES:
Anti-SARS-CoV2 seroprevalence in asymptomatic individuals at Day 0 | At enrollment (Day 0)
  Anti-SARS-Cov2 seroprevalence measured in serum samples collected at Day 0.
Anti-SARS-CoV2 seroprevalence in asymptomatic individuals at Day 21 | At Day 21
  Anti-SARS-Cov2 seroprevalence measured in serum samples collected at Day 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instuction des Armées Percy, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided